CLINICAL TRIAL: NCT00798356
Title: The Effect of Yoga on Arrhythmia Burden and Quality of Life in Patients With Paroxysmal Atrial Fibrillation
Brief Title: Yoga on Arrhythmia Burden and Quality of Life in Paroxysmal Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dhanunjaya Lakkireddy, MD, FACC (Other)
Responsible Party: Sponsor-Investigator, Dhanunjaya Lakkireddy, MD, FACC, Associate Professor of Medicine, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 11067
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation, yoga
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Yoga training
  Interventions: Other: Yoga training

INTERVENTIONS:
Other: Yoga training — Yoga training for 12 weeks

SUMMARY:
Studies in the past have shown that yoga could relieve stress which is the most common trigger for recurrent episodes of atrial fibrillation. Breathing exercises in yoga are found to influence the autonomic nervous system (particularly parasympathetic) and thus reduce palpitations. This study hypothesizes that patients with atrial fibrillation might benefit by practicing yoga. Yoga may also help to better control heart rate and rhythm when used in combination with usual medical management.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with paroxysmal atrial fibrillation ages 25-80

Exclusion Criteria:

* Advanced malignancy or severe co-morbid conditions such as severe heart failure and with life expectancy less than 1 year
* Pregnant women
* Unmedicated or uncontrolled high blood pressure
* A past history of pneumothorax
* Severe cervical spondylitis and cervical, thoracic or lumbar disc prolapse
* Carotid stenosis
* History of psychosis or substance abuse
* History of epilepsy
* Glaucoma
* History of total hip replacement
* Ablation within 3 months of the start date of study
* Patients who have not seen a cardiovascular physician in the last year

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2008-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
frequency and duration of atrial fibrillation episodes | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Lakkireddy D, Atkins D, Pillarisetti J, Ryschon K, Bommana S, Drisko J, Vanga S, Dawn B. Effect of yoga on arrhythmia burden, anxiety, depression, and quality of life in paroxysmal atrial fibrillation: the YOGA My Heart Study. J Am Coll Cardiol. 2013 Mar 19;61(11):1177-82. doi: 10.1016/j.jacc.2012.11.060. Epub 2013 Jan 30. PMID 23375926